CLINICAL TRIAL: NCT01937780
Title: Anal Cancer Radiotherapy - Prospective Study of Treatment Outcome, Patient-Reported Outcomes, Utility of Imaging and Biomarkers, and Cancer Survivorship
Brief Title: Anal Cancer Radiotherapy Study
Acronym: ANCARAD
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Grønlie Guren, MD PhD, Oslo University Hospital
Other Study IDs: 2012/2274
Record Dates: First submitted 2013-08-28; First posted 2013-09-10 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective study of patients receiving radiotherapy or chemoradiotherapy for anal cancer. Treatment effect in terms of survival and local recurrence will be analyzed. The utility of PET-CT and MRI for radiotherapy and for prediction of treatment effect will be investigated. Molecular and genetic markers in tumor and blood will be analyzed for prognostic and predictive effects. Patient-reported outcomes, such as faecal incontinence, sexual dysfunction and quality of life will be assessed. A structured intervention program for management of late effects will be evaluated. Symptom relief of palliative radiotherapy will be investigated. The main purpose of the study is to increase the knowledge of anal cancer treatment, improve treatment results, and improve anal cancer survivor care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified anal squamous cell carcinoma
* Radiotherapy or chemoradiotherapy planned
* ECOG performance status 0-2
* >= 18 years of age
* Signed informed consent and expected cooperation of the patients for treatment and follow up

Exclusion Criteria:

- Cognitive or physical condition resulting in inability to sign informed consent or cooperation during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anal cancer to be treated with radiotherapy or chemoradiotherapy
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-10-04 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
Prediction of local recurrence | 2 years
Biomarker ability to predict local recurrence rate | 5 years
  Substudy will analyze biomarkers in tissue/blood that may predict poor radiotherapy response or local recurrence.
Improvement of faecal incontinence | 5 years
Pain relief of palliative radiotherapy | 5 years
  Substudy will prospectively evaluate relief of pain and other symptoms of anal cancer after completion of palliative radiotherapy.

OTHER OUTCOMES:
Tumor regression | 5 years
PET and MRI prediction of local tumor control | 5 years
  Substudy will analyze PET and MRI at baseline and during treatment, for the ability to predict poor radiotherapy response or local recurrence rate.
To identify biomarkers predictive of treatment response or late effects | 5 years
Prevalence and severity of late effects in follow-up; fatigue, faecal incontinence, sexual dysfunction, health-related quality of life. Effect of intervention. | 5 years
Duration of symptom relief of palliative radiotherapy | 5 years
Local recurrence rate | 5 years
Disease-free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marianne G Guren, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway